CLINICAL TRIAL: NCT03153150
Title: Start or STop Anticoagulants Randomised Trial (SoSTART) After Spontaneous Intracranial Haemorrhage
Brief Title: Start or STop Anticoagulants Randomised Trial (SoSTART)
Acronym: SoSTART
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: SoSTART2016; 2016-004121-16 (EudraCT Number)
Record Dates: First submitted 2017-05-10; First posted 2017-05-15 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2021-05

CONDITIONS: Intracranial Hemorrhages; Intracranial Hemorrhage, Hypertensive; Subarachnoid Hemorrhage; Subdural Hematoma; Intraventricular Hemorrhage; Atrial Fibrillation; Atrial Flutter; Small Vessel Cerebrovascular Disease; Microhaemorrhage
Keywords: Oral anticoagulant; Factor Xa inhibitors; Direct thrombin inhibitor; Vitamin K antagonist; Antiplatelet drug
MeSH Terms: conditions — Intracranial Hemorrhages; Intracranial Hemorrhage, Hypertensive; Subarachnoid Hemorrhage; Hematoma, Subdural; Atrial Fibrillation; Atrial Flutter; Cerebral Small Vessel Diseases | interventions — apixaban; Rivaroxaban; edoxaban; Dabigatran; Acenocoumarol; Phenindione; Warfarin

STUDY DESIGN:
Intervention Model Description: 1:1 allocation of intervention: comparator, using a minimisation algorithm
Who Masked: Outcomes Assessor
Masking Description: PROBE design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Start oral anticoagulant (OAC) (Experimental): If the patient is randomized in this arm, an oral anticoagulant:
  * Factor Xa inhibitors: Apixaban or Rivaroxaban or Edoxaban or
  * Direct thrombin inhibitor: Dabigatran or
  * Vitamin K antagonists: Acenocoumarol or Phenindione or Warfarin chosen by the patient's physician before the randomisation, will be prescribed long-term (≥1 year) to the patient.
  Interventions: Drug: Apixaban; Drug: Rivaroxaban; Drug: Edoxaban; Drug: Dabigatran; Drug: Acenocoumarol; Drug: Phenindione; Drug: Warfarin
- Do not start oral anticoagulant (OAC) (No Intervention): If the patient is randomized in this arm, anticoagulant drugs will not be prescribed to the patient during the entire study period. The standard clinical practice without OAC may include:
  * antiplatelet drug(s) or
  * no antithrombotic drugs.

INTERVENTIONS:
Drug: Apixaban — The participant will be allocated to start this oral anticoagulant drug, if the participant's doctor indicated it before randomisation.
  Other Names: Eliquis
  Arms: Start oral anticoagulant (OAC)
Drug: Rivaroxaban — The participant will be allocated to start this oral anticoagulant drug, if the participant's doctor indicated it before randomisation.
  Other Names: Xarelto
  Arms: Start oral anticoagulant (OAC)
Drug: Edoxaban — The participant will be allocated to start this oral anticoagulant drug, if the participant's doctor indicated it before randomisation.
  Other Names: Lixiana
  Arms: Start oral anticoagulant (OAC)
Drug: Dabigatran — The participant will be allocated to start this oral anticoagulant drug, if the participant's doctor indicated it before randomisation.
  Other Names: Pradaxa
  Arms: Start oral anticoagulant (OAC)
Drug: Acenocoumarol — The participant will be allocated to start this oral anticoagulant drug, if the participant's doctor indicated it before randomisation.
  Other Names: Sinthrome
  Arms: Start oral anticoagulant (OAC)
Drug: Phenindione — The participant will be allocated to start this oral anticoagulant drug, if the participant's doctor indicated it before randomisation.
  Other Names: Dindevan
  Arms: Start oral anticoagulant (OAC)
Drug: Warfarin — The participant will be allocated to start this oral anticoagulant drug, if the participant's doctor indicated it before randomisation.
  Other Names: Marevan; Coumadin
  Arms: Start oral anticoagulant (OAC)

SUMMARY:
Primary research question: For adults surviving spontaneous (non-traumatic) symptomatic intracranial haemorrhage with persistent/paroxysmal atrial fibrillation/flutter (AF), does starting full treatment dose oral anticoagulation (OAC) result in a beneficial net reduction of all serious vascular events compared with not starting OAC?

Trial design: Investigator-led, multicentre, randomised, open, assessor-masked, parallel group, clinical trial of investigational medicinal product (CTIMP) prescribing strategies. Investigators plan for a pilot phase, followed by a safety phase.

DETAILED DESCRIPTION:
Bleeding within the skull, also known as brain haemorrhage, affects 3 million people in the world each year.

One in five people who survive brain haemorrhage have an irregular heart rhythm called 'atrial fibrillation', which puts them at risk of stroke and other blood clots.

Blood-thinning medicines, known as 'anticoagulant' drugs, are used in everyday clinical practice to protect people with atrial fibrillation from developing blood clots. However, these drugs also increase the risk of bleeding and are usually stopped when the brain haemorrhage occurs.

But when patients recover from brain haemorrhage, they and their doctors are often uncertain about whether to start or stop these drugs to prevent further clots occurring, or whether to avoid them in case they increase the risk of brain haemorrhage happening again.

Investigators want to find out whether starting or not starting an anticoagulant drugs is better for those patients.

A network of hospital doctors, nurses, and other staff will identify people who survive brain haemorrhage and have atrial fibrillation. If a patient and their doctor are uncertain about whether to start an anticoagulant drug, they may invite the patient to participate.

In the pilot phase, investigators aim to recruit at least 60 participants to determine the feasibility of recruiting the target sample size of at least 190 participants in the safety phase of the trial.

Investigators will follow-up all participants for at least one year to determine whether prescribing an anticoagulant drug reduces the occurrence of all serious vascular events like heart attack, stroke compared with a policy of avoiding oral anticoagulant.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age ≥18 years
2. Symptomatic intracranial haemorrhage (i.e. intracerebral haemorrhage, non-aneurysmal subarachnoid haemorrhage,intraventricular haemorrhage, or subduralhaemorrhage)

   * Not attributable to a known underlying intracranial aneurysm, arteriovenous malformation, cerebral cavernous malformation, dural arteriovenous fistula, intracranial venous thrombosis
   * Not attributable to known head injury, based on:
   * a history from the patient/witness of spontaneous symptom onset without preceding head trauma (head trauma occurring after symptom onset is permissible)
   * brain imaging appearances consistent with spontaneous intracranial haemorrhage (which may be accompanied by the brain/bone/soft tissue appearances of trauma occurring subsequently)
3. Atrial fibrillation/flutter (persistent or paroxysmal) with a CHA2DS2-VASc score ≥2
4. If included in the brain magnetic resonance imaging (MRI) sub-study, the scan must be done after symptomatic intracranial haemorrhage and before randomisation

Exclusion Criteria:

1. Symptomatic intracranial haemorrhage within the last 24 hours (when the risk of haemorrhage expansion/growth is greatest)
2. Symptomatic intracranial haemorrhage is exclusively due to trauma or haemorrhagic transformation of ischaemic stroke
3. Prosthetic mechanical heart valve or severe (haemodynamically significant) native valve disease
4. Left atrial appendage occlusion for prevention of systemic embolism in AF done in the past, or intended to be performed
5. Intention to start antiplatelet drug(s) if randomised to start full dose OAC
6. Intention to start OAC or parenteral anticoagulation
7. Intention to implement the allocated treatment strategy for <1 year
8. Patient or their doctor is certain about whether to start or avoid full dose OAC
9. Brain imaging that first diagnosed the intracranial haemorrhage is not available
10. Patient is not registered with a general practitioner
11. Patient is pregnant, breastfeeding, or of childbearing age and not taking contraception
12. Patient and carer unable to understand spoken or written English
13. Contraindications to any of the IMPs, other than recent intracranial haemorrhage
14. Contraindication to MRI (brain MRI sub-study)
15. Life expectancy less than one year
16. Previously randomised in SoSTART

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2018-03-28 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

PRIMARY OUTCOMES:
The number of participants recruited per site per month (in the pilot phase of the trial) | 1 year after trial initiation
  The rate of recruiting up to 60 participants to determine the feasibility of recruiting the target sample size in the main phase of the trial in an acceptable timescale.
Recurrent symptomatic spontaneous intracranial haemorrhage (in the safety phase of the trial) | 1 year after randomisation
  ~60 hospital sites will recruit at least 190 participants to determine whether the risk of recurrent symptomatic intracranial haemorrhage is sufficiently low (non-inferior) to justify a definitive trial.

SECONDARY OUTCOMES:
The proportions of all eligible patients recorded on screening logs who are recruited, unsuitable, or decline to participate (in the pilot phase of the trial) | 1 year after randomisation
  The acceptability of the trial protocol to investigators and patients.

OTHER OUTCOMES:
The number of Symptomatic serious vascular events: (in the safety phase of the trial) | 1 year after randomisation
  • All symptomatic serious vascular events (i.e. major adverse cardiac or cerebrovascular events [MACCE]) including: non-fatal (i.e. not followed by death within 30 days of onset) myocardial infarction; stroke (i.e. ischaemic, haemorrhagic, unknown sub-type) or spontaneous subdural haemorrhage; or death from a vascular cause (i.e. haemorrhagic or ischaemic events followed by death within 30 days), sudden death, or death of an unknown cause.
The number of Individual symptomatic vascular events: (in the safety phase of the trial) | 1 year after randomisation
  * Major haemorrhagic events (Bleeding Academic Research Consortium types 3-5)
    * Recurrent symptomatic spontaneous intracranial haemorrhage
    * Extracranial haemorrhage
  * Symptomatic ischaemic events
    * ischaemic stroke
    * myocardial infarction
    * peripheral arterial occlusion
    * mesenteric ischaemia
    * central retinal arterial occlusion
    * deep vein thrombosis
    * pulmonary embolism
    * cardiac death with symptoms suggestive of myocardial ischaemia (type 3),or evidence of arrhythmia
  * Revascularisation procedures (carotid, coronary, or peripheral arterial)
  * Symptomatic stroke of uncertain sub-type
    * Non-fatal stroke, with brain imaging performed too late to distinguish haemorrhage from infarction
    * Rapidly fatal stroke, but without radiographic or pathological confirmation
Annual ratings of participant dependence completed by participant, their carer or nominated contact, or healthcare provider (e.g. general practitioner): | 1 year after randomisation
  • Simplified modified Rankin Scale
Ratings of participant quality of life completed by participant, their carer or or nominated contact | Randomisation and 1 year after randomisation
  • The 5-level EQ-5D version (EQ-5D-5L) of the EuroQol

CONTACTS AND LOCATIONS:
Overall Officials: Rustam Al-Shahi Salman, MA PhD FRCP, Principal Investigator — University of Edinburgh
Locations (67):
- United Kingdom (67):
  - Edinburgh Royal Infirmary, Edinburgh, Midlothian
  - Aberdeen Royal Infirmary, Aberdeen
  - Nevill Hall Hospital, Abergavenny
  - Monklands Hospital, Airdrie
  - Barnet Hospital, Barnet
  - Royal United Hospital, Bath
  - Heartlands Hospital, Birmingham
  - The Royal Bournemouth Hospital, Bournemouth
  - Bradford Royal Infirmary, Bradford
  - University Hospital Bristol, Bristol
  - Addenbrookes Hospital, Cambridge
  - University Hospital of Wales/ /University Hospital Llandough, Cardiff
  - Colchester General Hospital, Colchester
  - Derby Royal Hospital, Derby
  - University Hospital North Durham, Durham
  - South West Acute Hospital, Enniskillen
  - Royal Devon & Exeter Hospital, Exeter
  - Frimley Park Hospital, Frimley
  - Queen Elizabeth Hospital, Gateshead
  - Medway Maritime Hospital, Gillingham
  - Glasgow Royal Infirmary, Glasgow
  - Queen Elizabeth University Hospital, Glasgow
  - Gloucestershire Royal Hospital, Gloucester
  - Calderdale Royal Hospital, Halifax
  - Northwick Park, Harrow
  - Ystrad Mynach Hospital, Hengoed
  - Victoria Hospital Kirkcaldy, Kirkcaldy
  - Royal Lancaster Infirmary, Lancaster
  - Leeds General Infirmary, Leeds
  - Royal Liverpool and Broadgreen University Hospital, Liverpool
  - University Hospital Aintree, Liverpool
  - The Royal London Hospital, London
  - Homerton University Hospital, London
  - North Middlesex University Hospital, London
  - University College London Hospital, London
  - St Thomas Hospital, London
  - St.George's Hospital, London
  - Altnagelvin Hospital, Londonderry
  - Luton & Dunstable University Hospital, Luton
  - King's Mill Hospital, Mansfield
  - Arrowe Park Hospital, Metropolitan Borough of Wirral
  - James Cook University Hospital, Middlesbrough
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - Nottingham City Hospital, Nottingham
  - John Radcliffe Hospital, Oxford
  - Peterborough City Hospital, Peterborough
  - Poole Hospital, Poole
  - Royal Preston Hospital, Preston
  - Royal Berkshire Hospital, Reading
  - Queen' Hospital Romford, Romford
  - Salford Royal NHS Foundation Trust, Salford
  - Royal Hallamshire Hospital, Sheffield
  - Southampton General Hospital, Southampton
  - University Hospital of North Tees, Stockton-on-Tees
  - Royal Stoke University Hospital, Stoke-on-Trent
  - Sunderland Royal Hospital, Sunderland
  - Morriston Hospital, Swansea
  - The Princess Royal Hospital, Telford
  - Torbay District General Hospital, Torquay
  - Royal Cornwall Hospital, Truro
  - Hillingdon Hospital, Uxbridge
  - Pinderfields Hospital, Wakefield
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea
  - Royal Hampshire County Hospital, Winchester
  - New Cross Hospital, Wolverhampton
  - Yeovil District Hospital, Yeovil
  - York Hospital, York

IPD SHARING:
Plan to Share IPD: Yes
The Chief Investigator (Prof. Rustam Al-Shahi Salman) has established the Collaboration Of Controlled Randomised trials of Oral Antithrombotic drugs after intraCranial Haemorrhage (COCROACH) working towards a pre-planned individual patient data meta-analysis

REFERENCES:
- [Result] SoSTART Collaboration. Effects of oral anticoagulation for atrial fibrillation after spontaneous intracranial haemorrhage in the UK: a randomised, open-label, assessor-masked, pilot-phase, non-inferiority trial. Lancet Neurol. 2021 Oct;20(10):842-853. doi: 10.1016/S1474-4422(21)00264-7. Epub 2021 Sep 3. PMID 34487722
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520
- [Derived] Li L, Poon MTC, Samarasekera NE, Perry LA, Moullaali TJ, Rodrigues MA, Loan JJM, Stephen J, Lerpiniere C, Tuna MA, Gutnikov SA, Kuker W, Silver LE, Al-Shahi Salman R, Rothwell PM. Risks of recurrent stroke and all serious vascular events after spontaneous intracerebral haemorrhage: pooled analyses of two population-based studies. Lancet Neurol. 2021 Jun;20(6):437-447. doi: 10.1016/S1474-4422(21)00075-2. PMID 34022170
- See also: Trial website — http://www.sostart.ed.ac.uk
- See also: Chief investigator details — http://www.rush.ed.ac.uk